CLINICAL TRIAL: NCT03483324
Title: A Phase 1 Open-Label, Multi-Center Trial of AB-110 in Adults With Hematologic Malignancies Undergoing Cord
Brief Title: Trial of AB-110 in Adults With Hematologic Malignancies Undergoing Cord Blood Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Angiocrine Bioscience (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-110-001
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia in Remission; Myelodysplastic Syndromes; Other Acute Leukemias
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — epithienamycin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Unmanipulated umbilical cord blood plus AB-110
  Interventions: Biological: Unmanipulated Umbilical Cord Blood (UCB); Biological: AB-110

INTERVENTIONS:
Biological: Unmanipulated Umbilical Cord Blood (UCB) — Human leukocyte antigen (HLA) matched umbilical cord blood
Biological: AB-110 — Expanded cord blood stem cells and engineered human endothelial cells

SUMMARY:
A phase 1b, open label, multi-center trial of AB-110 in adults with hematologic malignancies, including acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), and myelodysplasia (MDS) undergoing cord blood transplantation. Subjects will receive unmanipulated cord blood (UCB) and AB-110 expanded CD34 enriched hematopoietic progenitor cells (HSPC).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received some immunosuppressive chemotherapy in the preceding 3 months.
* Acute myelogenous leukemia (AML):

  1. Complete first remission (CR1) at high risk for relapse
  2. Complete second remission (CR2).
  3. No documented myelofibrosis at screening marrow biopsy
* Acute lymphoblastic leukemia (ALL):

  1. Complete first remission (CR1) at high risk for relapse
  2. Complete second remission (CR2).
* Other acute leukemias that are of ambiguous lineage or of other types
* Any acute leukemia with marrow aplasia or without adequate count recovery.
* Myelodysplastic Syndrome (MDS)
* Karnofsky score > 70 %.
* Calculated creatinine clearance > 60 ml/min.
* Bilirubin < 1.5 mg/dL, ALT < 3 x upper limit of normal
* Pulmonary function (FVC, FEV1 and corrected DLCO) > 50% predicted.
* Left ventricular ejection fraction > 50%.
* Albumin > 3.0 g/dL.
* Negative antiviral serology:
* Negative human immunodeficiency virus (HIV) antibody.
* Negative human T-lymphotropic virus (HTLV)-1 and 2 antibodies.
* Negative hepatitis B surface antigen (HBsAg) and undetectable hepatitis B virus (HBV) DNA
* Negative hepatitis C virus (HCV) antibody or negative HCV ribonucleic acid (RNA)
* For female subjects of childbearing potential:

  1. A negative serum pregnancy test
  2. Willing to use contraception throughout the study period.
* Male subjects must be willing to use a recommended method of contraception throughout the study period, and to refrain from sperm donation throughout the study period.
* Two appropriate CB units identified for the subject.
* In the judgment of the investigator, participation in the protocol offers an acceptable benefit-to-risk ratio when considering current disease status, medical condition, and the potential benefits and risks of alternative treatments for the subject's cancer.
* Willingness and ability to comply with scheduled visits, drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions.
* Evidence of a signed informed written consent

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Current active, uncontrolled bacterial, viral, or fungal infection
* Prior allogeneic or autologous HCT at any time.
* Active malignancy other than the one for which AB-110 transplant is being performed within 12 months of enrollment.
* Any identified and available 10/10 HLA-matched related donor or 10/10 HLA-matched unrelated donor.
* Have evidence of recipient donor specific anti-HLA antibodies.
* Active central nervous system (CNS) disease at time of screening.
* Documented allergy to DMSO, mouse or bovine proteins, or iron.
* Subject has other conditions that in the opinion of the investigator would place the subject at increased risk for toxicity by participation in the study.
* Psychiatric condition making the patient unlikely to comply with protocol therapy, required tests and follow-up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events grade 4 or grade 5 as assessed by CTCAEv4 | 24 hours
Graft failure defined as survival to day 42 without absolute neutrophil count greater than or equal to 500/mm3 | 42 days

SECONDARY OUTCOMES:
Time to neutrophil engraftment | 42 days
Cumulative incidence of sustained donor-derived neutrophil engraftment | 42 days
Cumulative incidence of sustained donor-derived neutrophil engraftment | 100 days
Cumulative incidence of sustained donor-derived neutrophil engraftment | 180 days
Incidence of engraftment syndrome | 28 days
Cumulative incidence of graft failure | 43 days
Cumulative incidence of graft failure | 180 days
Presence of post-transplant phenotype in hematopoietic cells of donor origin | 180 days
Cumulative incidence of grade II - IV acute graft versus host disease (aGVHD) | 100 days
Cumulative incidence of grade II - IV acute graft versus host disease (GVHD) | 180 days
Cumulative incidence of chronic GVHD | 100 days
Cumulative incidence of chronic GVHD | 180 days
Time to lymphoid recovery | 180 days
Cumulative incidence of transplant related mortality (TRM) | 100 days
Cumulative incidence of transplant related mortality (TRM) | 180 days
Overall survival (OS) | 100 days
Overall survival (OS) | 180 days
Disease Free Survival (DFS) | 100 days
Disease Free Survival (DFS) | 180 days

OTHER OUTCOMES:
Late onset acute GVHD | 720 days
Chronic GVHD | 720 days
Quantitative recovery of T-cells and subsets | 1 year
Quantitative recovery of T-cells and subsets | 2 years
Transplant Related Mortality | 1 year
Transplant Related Mortality | 2 years
Recurrence of malignancy | 1 year
Recurrence of malignancy | 2 years
Overall survival | 1 year
Overall survival | 2 years
Disease free survival | 1 year
Disease free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Finnegan, MD, Study Director — Angiocrine Bioscience
Locations (3):
- United States (3):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of Colorado Cancer Center University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No